CLINICAL TRIAL: NCT06921330
Title: The Effect of White Cover and Massage Application on Bilirubin Levels and Duration of Phototherapy in Newborns With ABO Incompatibility Receiving Phototherapy
Brief Title: White Cover & Massage Effects on Bilirubin and Phototherapy in ABO-Incompatible Newborns
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Zeynep ÇİFTCİ DEMİRTAŞ, Midwife, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-77192459-050.99-382574
Record Dates: First submitted 2025-03-28; First posted 2025-04-10 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Newborn Jaundice; Hyperbilirubinemia, Neonatal; ABO Incompatibility; Newborn Massage; Phototherapy; White Cover
Keywords: ABO incompatibility; newborn; phototherapy; White cover; massage; Hyperbilirubinemia
MeSH Terms: conditions — Jaundice, Neonatal; Hyperbilirubinemia, Neonatal; Hyperbilirubinemia | interventions — Massage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): 1. During phototherapy, the phototherapy devices of term newborns with abo incompatibility will be covered with white cover.
  2. During phototherapy, infant massage including facial massage, chest massage, arm massage, abdominal massage and leg massage will be applied to term newborns twice a day for 15 minutes each session with an interval of 6 hours.
  Interventions: Other: white cover-newborn massage
- control group (No Intervention): The hospital's clinical routine will be applied to the newborns in the control group.

INTERVENTIONS:
Other: white cover-newborn massage — A white cover will be covered over the incubator during phototherapy. Baby massage will be applied during phototherapy.
  Other Names: white cover and massage
  Arms: intervention group

SUMMARY:
This study aims to examine the effect of white cover and massage application on bilirubin levels and phototherapy duration in newborns with ABO incompatibility receiving phototherapy.

DETAILED DESCRIPTION:
Hyperbilirubinemia is a common problem seen in the neonatal period characterized by yellow staining of the skin and sclera, causing an increase in total serum bilirubin >5 mg/dl. Neonatal jaundice is observed in 60% of term newborns and 80% of preterm newborns. Hyperbilirubinemia is usually physiologic and disappears within a few days. If jaundice becomes severe and pathologic hyperbilirubinemia occurs, it can lead to kernicterus (bilirubin accumulation in parts of the brain) or death.Therefore, any infant with hyperbilirubinemia with elevated serum bilirubin levels requires serious attention and treatment.

ABO incompatibility is a cause of indirect hyperbilirubinemia leading to pathologic jaundice. Newborns with ABO incompatibility tend to have higher bilirubin levels due to impaired bilirubin excretion during the neonatal period. ABO incompatibility is observed in approximately 25% of mother-infant pairs. ABO incompatibility may develop when the mother's blood type is O and the baby's blood type is A or B. In ABO incompatibility, maternal anti-A or anti-B antibodies cross the placenta and bind to A/B antigens on the surface of fetal erythrocytes. Antibody-coated erythrocytes are destroyed in the reticuloendothelial system. Bilirubin increases as a result of heme catabolism that is released with the destruction of erythrocytes, and this is reflected in the clinic as neonatal jaundice. In the presence of ABO incompatibility, early screening and close follow-up of newborns in terms of development of hyperbilirubinemia is very important. Traditional treatment modalities for jaundice due to ABO incompatibility are phototherapy and exchange transfusion.

The primary treatment of neonatal jaundice is phototherapy. The efficacy of phototherapy depends on the phototherapy light source, light intensity, the distance between the phototherapy light and the newborn, and the body surface area exposed to light. Phototherapy has potential side effects such as hyperthermia, dehydration, diarrhea, bronze baby syndrome and skin burns in newborns. Therefore, the use of phototherapy should be minimized and solutions should be found to shorten the duration of phototherapy. To increase the effectiveness of phototherapy treatment, a reflective material can be added to the phototherapy. White fabric that can be used as a reflector can reflect the scattered phototherapy light. When fabrics made of reflective materials are hung on the phototherapy device, they can capture light that may be scattered from the baby to the environment and reflect the light back to the baby. The white fabric can increase the irradiance and thus increase bilirubin conversion. Bilirubin is excreted from the body through feces. Removal of bilirubin from the body reduces jaundice. Massage decreases bilirubin levels by increasing the frequency of bowel movements in newborn babies.

ELIGIBILITY:
Inclusion Criteria:

* Abo-Incompatibility term babies with a gestational age between 37-42 weeks,
* Does not have a respiratory, cardiovascular, gastrointestinal or neurological disorder or syndrome that would prevent or complicate oral feeding,
* Birth weight of 2500 g and above,
* With phototherapy indication,
* Do not have any health problems other than neonatal jaundice detected in the prenatal period,
* Those with a stable health condition,
* Orally fed,
* No clinical signs of dehydration,
* Do not have any skin problems that would prevent baby massage,
* Newborns with written and verbal informed consent from their families will be included in the study.

Exclusion Criteria:

* Premature,
* Those with congenital malformations,
* Those with hyperbilirubinemia requiring exchange transfusion,
* Those with Rh hemolytic disease,
* Having a positive culture test (sepsis),
* Those with glucose-6-phosphate dehydrogenase (G6PD) deficiency,
* Birth weight below 2500 grams,
* Those who were referred to another center during the research,
* Discharged early,
* Unexpected complications developed during the research,
* Bronze child syndrome occurs during phototherapy,
* Newborns who develop a pathology that will prevent or complicate oral feeding will not be included in the study.

Ages: 12 Hours to 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-05 (Estimated)

PRIMARY OUTCOMES:
Change in bilirubin level | From immediately before initiation of phototherapy to immediately after termination of phototherapy
  Capillary bilirubin levels will be measured immediately before the initiation of phototherapy and immediately after the termination of phototherapy. The change in capillary bilirubin levels will be calculated and reported.The unit of measure for bilirubin levels will be milligrams per deciliter (mg/dL).
Duration of phototherapy | From initiation to termination of phototherapy
  The total duration of phototherapy required until bilirubin levels decreased below the treatment threshold will be recorded.The unit of measure for the duration of phototherapy is hours.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep ze ÇİFTCİ DEMİRTAŞ, 1, Principal Investigator — midwife
Locations (1):
- Karabük Eğitim Ve Araştırma Hastanesi, Karabük, Karabük Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No